CLINICAL TRIAL: NCT02122315
Title: EFFECTIVENESS OF THE INCLUSION OF TRIGGER POINT DRY NEEDLING INTO A MULTIMODAL PHYSICAL THERAPY PROGRAM FOR POST-OPERATIVE SHOULDER PAIN
Brief Title: Dry Needling in Post-operative Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: César Fernández-de-las-Peñas (Other)
Responsible Party: Sponsor-Investigator, César Fernández-de-las-Peñas, Head Division, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP13-060
Record Dates: First submitted 2014-04-19; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Proximal Humeral Fracture Fixated With PHILOS© Plate; Rotator Cuff Tear Surgical Repair
MeSH Terms: interventions — Physical Therapy Modalities; Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical therapy plus dry needling (Experimental): Best-evidence physical therapy intervention in addition to a single session of TrP-DN targeted to active TrPs in the neck-shoulder muscles.
  Interventions: Other: Physical therapy plus dry needling
- Physical therapy (Active Comparator): Best-evidence physical therapy intervention
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Physical therapy plus dry needling — Best-evidence physical therapy intervention in addition to a single session of TrP-DN targeted to active TrPs in the neck-shoulder muscles
  Arms: Physical therapy plus dry needling
Other: Physical therapy — Best-evidence physical therapy intervention
  Arms: Physical therapy

SUMMARY:
Fractures of the proximal humerus account for between 5% and 8% off all reported fractures. Post-operative shoulder pain is highly frequent. Due to either surgical procedure, soft tissues surrounding the shoulder area can be damaged. The purpose of the current clinical trial was to compare the effects of physiotherapy versus physiotherapy plus TrP-DN on pain and function in patients who exhibit post-operative shoulder pain after a PHILOS procedure for proximal humeral fixation or rotator cuff tear repair.

ELIGIBILITY:
Inclusion Criteria:

* proximal humeral fracture
* rotator cuff tear
* open reduction and internal fixation with PHILOS© plate (Synthes, Switzerland)
* rotator cuff tear repair
* post-operative shoulder pain
* active TrPs in the neck-shoulder muscles

Exclusion Criteria:

* no active TrPs
* multiple fracture
* previous surgery
* cervical radiculopathy or myelopathy
* diagnosis of fibromialgia
* having undergone any physical therapy intervention in the year before the surgery
* fear of needles
* any contraindication for dry needling

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Changes in Constant-Murley score before and after the intervention | Baseline and one week after the intervention
  The Constant-Murley score is a 100-point scoring system that is divided into 4 main sub-scales: pain (15 points); activities of daily living (20 points); range of motion (40 points); and strength (25 points). Higher score represents better function

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Fernández-de-las-Peñas, PhD, Study Chair — Universidad Rey Juan Carlos
Locations (1):
- Jose Luis Arias Buría, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196